CLINICAL TRIAL: NCT02707081
Title: Efficacy of Intraperitoneal Versus Intravenous Lidocaine for Postcesarean Pain Relief
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Walid Anwar Murad, Assistant Professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Benha 121
Record Dates: First submitted 2016-03-04; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Postcesarean Pain Relief
MeSH Terms: interventions — Sodium Chloride; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo control group (Placebo Comparator): Saline was given both intraperitoneally and intravenously during caesarean section
  Interventions: Drug: Intravenous normal saline; Drug: Intraperitoneal normal saline
- Intraperitoneal instillation group (Active Comparator): Patients received 1.75 ml/kg of 0.2% lidocaine (3.5mg/kg) with parietal peritoneal closure with intravenous normal saline in a volume equivalent to that used in intravenous lidocaine group as placebo to ensure blinding.
  Interventions: Drug: Intravenous normal saline; Drug: Intraperitoneal Lidocaine
- Intravenous injection group (Active Comparator): Patients received 1.5mg/kg of intravenous 1% lidocaine as bolus dose at induction and 2mg/kg/hour as continuous infusion of intravenous lidocaine until one hour after surgery and 100 ml of saline intraperitoneally as placebo to ensure blinding
  Interventions: Drug: Intraperitoneal normal saline; Drug: Intravenous Lidocaine

INTERVENTIONS:
Drug: Intravenous normal saline — Normal saline in a volume equivalent to that used in intravenous lidocaine group
  Other Names: IV Saline
  Arms: Intraperitoneal instillation group; Placebo control group
Drug: Intraperitoneal normal saline — Patients received 00 ml of saline intraperitoneally
  Other Names: IP Saline
  Arms: Intravenous injection group; Placebo control group
Drug: Intraperitoneal Lidocaine — Patients received 1.75 ml/kg of 0.2% lidocaine (3.5mg/kg) with parietal peritoneal closure.
  Other Names: IP Lidocaine
  Arms: Intraperitoneal instillation group
Drug: Intravenous Lidocaine — Patients received 1.5mg/kg of intravenous 1% lidocaine as bolus dose at induction and 2mg/kg/hour as continuous infusion of intravenous lidocaine until one hour after surgery.
  Other Names: IV Lidocaine
  Arms: Intravenous injection group

SUMMARY:
Objective: To evaluate intraperitoneal (IP) lidocaine administration and intravenous (IV) lidocaine infusion for postoperative pain control after cesarean section.

Study design: prospective randomized, double-blind, placebo-controlled study. Patients and methods: Initially, 165 pregnant full-term females, indicated to be underwent elective cesarean delivery for various indications were randomized equally to either group C (control, IP and IV saline), group IP (intraperitoneal lidocaine administration), or group IV (intravenous lidocaine infusion).Five patients were excluded from each group for various reasons. The outcome measures were postoperative pain scoring, total pethidine consumption and the need for postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy, more than or equal completed 37 gestational weeks, indicated to undergo elective cesarean delivery for various indications

Exclusion Criteria:

* extreme of age (below 18 or above 40 year), uncooperative patients, women under spinal anesthesia, previous abdominal scars, including previous cesarean or myomectomy, multiple gestation, BMI >35 kg/m², chorioamnionitis, hypersensitivity or contraindications to lidocaine, bronchial asthma, bleeding diathesis, pregnancy induced-hypertension, liver or kidney diseases, diabetes mellitus, and patients with psychological disturbance, or any form of chronic pain before or during pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scoring (number) | First 24 hours postoperative

SECONDARY OUTCOMES:
The need for rescue postoperative analgesia. | First 24 hours postoperative
Total pethidine consumption in 24 hours (mg) | First 24 hours postoperative
The time to bowel sounds, hours | First 3 days postoperative
The time to start regular diet, days | First 3 days postoperative
Duration of hospital stay , days | First 3 days postoperative
Any reported side effects | First 3 days postoperative